CLINICAL TRIAL: NCT02484222
Title: Fentanyl Test Results and Its Association With Morphine Requirements in Children With Obstructive Sleep Apnea Syndrome After Adenotonsillectomy
Brief Title: Fentanyl Test in Children's Adenotonsillectomy
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xuan Wang, Doctor, Children's Hospital of Fudan University
Other Study IDs: FTCA-01
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: adenotonsillectomy; fentanyl
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fentanyl — Before the end of the procedure, spontaneous respiratory was recovered. All the patients were given 1 mcg/kg fentanyl i.v. after the end of the procedure.
  Other Names: Fentanyl test

SUMMARY:
The purpose of this study is to discuss the relationship between the result of fentanyl test and required dosage of morphine for children with OSAS after adenotonsillectomy；and to evaluate the ability of predicting requested dosage of morphine postoperatively.

DETAILED DESCRIPTION:
All the patients were intubated. Sevoflurane was used for maintenance without any opioids. Before the end of the procedure, spontaneous respiratory was recovered. All the patients were given 1 mcg/kg fentanyl i.v. after the end of the procedure. The positive result was defined as spontaneous respiratory rate decreased more than 50%, the others were defined as negative result. All the patients were given morphine for pain relief according to our protocol after extubation.

ELIGIBILITY:
Inclusion Criteria:meet all of the following

1. the American society of anesthesiologists (ASA) class Ⅰ ~ Ⅱ
2. the age of 3 ~ 7 years old
3. children who underwent selective adenotonsillectomy.

Exclusion Criteria:meet anyone of the following

1. craniofacial malformations
2. mental retardation
3. BMI > 22 kg/m2
4. a history of bronchial asthma
5. a recent history of opioid use.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who were diagnosed with Obstructive Sleep Apnea Syndrome(OSAS) by electronic nasopharyngoscope and underwent selective adenotonsillectomy
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Wang, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Chilren's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li YH, Wang X, Zhou ZJ, Zhuang PJ. Association between fentanyl test results and rescue morphine requirements in children after adenotonsillectomy. J Anesth. 2018 Feb;32(1):77-81. doi: 10.1007/s00540-017-2433-0. Epub 2017 Nov 21. PMID 29164334

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children at age of 3 - 7 years with OSAS,The exclusion criteria were craniofacial deformities, mental retardation, BMI > 22 kg/m², a history of bronchial asthma, and a recent history of opioid use.
Groups:
- The Result of Fentanyl Test: The children were divided by the breath decreasing rates-with 50% decreasing rate of breath were positive result, and the rest were negative.
Period: Overall Study
Arm/Group | The Result of Fentanyl Test
Started | 80
Completed | 77
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | The Result of Fentanyl Test
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5.2 [3.9 to 6.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  China | 80

OUTCOME MEASURES:

1. Primary Outcome: Rescue Morphine Requirement
Time Frame: average 1 hour from extubation
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | The Result of Fentanyl Test
Number analyzed (Participants) | 77
mg | 30 [20 to 40]

2. Secondary Outcome: Post-operative Nausea and Vomiting
Time Frame: average 1 hour from extubation
Measure: Count of Participants; unit: Participants
Groups:
- Nausea and Vomiting: post-operative nausea and vomiting
Arm/Group | Nausea and Vomiting
Number analyzed (Participants) | 77
Participants | 13

3. Secondary Outcome: Number of Participants With Pulse Oxygen Saturation Less Than 95 Percent
Time Frame: average 1 hour from extubation
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Pulse Oxygen Saturation Less Than: Number of Participants with Pulse Oxygen Saturation Less Than 95 Percent
Arm/Group | Number of Participants With Pulse Oxygen Saturation Less Than
Number analyzed (Participants) | 77
Participants | 7

4. Post Hoc Outcome: Number of Participants Who Were Light Consumers of Morphine as Identified by the Fentanyl Test
Description: The number of participants who were light consumers of morphine as identified by the Fentanyl Test，we want to know the accurate of the test.The light consumers are the children of who used total morphine <50 μg/kg.
Time Frame: average 1 hour from extubation
Measure: Count of Participants; unit: Participants
Arm/Group | The Result of Fentanyl Test
Number analyzed (Participants) | 77
Participants | 47

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Post-operative Nausea/vomiting (PONV) and other adverse events, such as airway obstruction, laryngospasm.
Arm/Group | The Result of Fentanyl Test
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 13/77
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Result of Fentanyl Test (N=77)
vomiting (General disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes